CLINICAL TRIAL: NCT00808548
Title: Exploring Stress and Coping Behaviors of the Major Carer Whose Children With Prader-Willi Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: shu chien, Taichung Veterans General Hospital
Other Study IDs: C08169
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Prader-Willi Syndrome
Keywords: stress; carer's experiences; Prader-willi syndrome; personal experiences
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lifestyle counseling
  Interventions: Other: counseling, emotional support; Other: emotional support

INTERVENTIONS:
Other: counseling, emotional support
Other: emotional support — emotional support during the interview
Other: emotional support — emotional supporting during the interview

SUMMARY:
Ask the 4 carers of children with Prader-willi syndrome to disclose their experiences and difficulties for searching better management and intervention

ELIGIBILITY:
Inclusion Criteria:

* a person who care and live with children with Prader-Willi syndrome

Exclusion Criteria:

* siblings or less-contact family
* teachers

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: a person who care and live with childre with Prader-Willi syndrome
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-02 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
experience | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan